CLINICAL TRIAL: NCT06179563
Title: Enhancing Patient Empowerment in Inflammatory Bowel Disease: The Role of On-Demand Telemonitoring
Brief Title: TOD-IBD: Empowering Patients On-Demand
Acronym: TOD-IBD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Collaborators: Jeroen Bosch Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: NL86106.100.24
Record Dates: First submitted 2023-12-05; First posted 2023-12-22 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases; Telemonitoring; Patient Empowerment; Self Efficacy
Keywords: Monitor IBD At Home; Fecal Calprotectin; On-Demand; Appropriate Care
MeSH Terms: conditions — Inflammatory Bowel Diseases; Patient Participation

STUDY DESIGN:
Intervention Model Description: Pragmatic, multicentre, randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard telemonitoring (No Intervention): Patients will be monitored according to a fixed telemonitoring schedule at their treating hospitals, based on the patient's medication type and in adherence to national and international guidelines.
- On-Demand Telemonitoring (Experimental): Patients will have the flexibility to use the telemonitoring application at their own discretion
  Interventions: Other: On-Demand Telemonitoring

INTERVENTIONS:
Other: On-Demand Telemonitoring — Patients assigned to the on-demand intervention group do not have to use the app at set time intervals but will be asked to use the app at their own discretion, in case of symptoms. This implies that patients have full control over their monitoring activities. Patients have the option to reach out to the hospital whenever they feel the need.
  Arms: On-Demand Telemonitoring

SUMMARY:
Crohn's disease and Ulcerative Colitis, collectively known as Inflammatory Bowel Disease (IBD), impose a significant burden on patients and healthcare systems due to their chronic nature and complex treatment. This study aims to assess the effectiveness and safety of on-demand telemonitoring, as opposed to standard fixed-schedule telemonitoring, in managing IBD. The primary objective is to evaluate the impact of on-demand telemonitoring on the number of persistent flares over 12 months. The study involves a multicenter randomized controlled trial comparing standard telemonitoring, which includes regular completion of the Monitor IBD At Home questionnaire and fecal calprotectin home tests, with on-demand telemonitoring where patients use the app based on their symptoms. The study population includes adult patients with stable remission on maintenance therapy. Disease activity, measured by unplanned healthcare contacts, is the primary outcome, while secondary outcomes encompass clinical and patient-reported disease activity, quality of life, self-efficacy, patient activation, total healthcare contacts, safety, and costs. Baseline characteristics include patient, disease, and socio-demographic factors. This innovative approach has the potential to enhance patient autonomy, satisfaction, and self-management, while reducing the overall burden on the healthcare system.

DETAILED DESCRIPTION:
Rationale: Crohn's disease and Ulcerative Colitis (Inflammatory Bowel Disease (IBD)) are chronic intestinal inflammations with significant impact on quality of life. Due to their chronic nature and complex treatment requiring regular outpatient appointments, IBD care puts a great burden on both the patient and the healthcare system. Appropriate care, as described in the Integrated Care Agreement published by the Dutch ministry of Health, is becoming increasingly important. Telemonitoring is a promising alternative to regular outpatient visits, with even evidence of improving the quality of care. We combined a clinical disease activity patient-reported outcome measure (the Monitor IBD At Home questionnaire) with a faecal calprotectin home test (SmarTest from Preventis) integrated in a new easy to use E-health application IBD Care Everywhere (IBD-CE) for IBD patients to determine disease activity at home.

In this study, we investigate whether using telemonitoring on-demand, according to individual needs, is equally effective and safe as telemonitoring based on a fixed schedule. This concept offers the opportunity to align the treatment of the disease more closely with the principles of appropriate care, which can result in improved patient autonomy, increased satisfaction, and enhanced self-management, while simultaneously reducing the burden on the healthcare system.

Objective: The primary objective is to assess the effect of on-demand telemonitoring for IBD patients on the number persistent flares for 12 months follow up.

Study design and intervention: This is a multicenter randomized controlled trial comparing on-demand telemonitoring with standard telemonitoring over a period of 12 months. Patients in the standard telemonitoring group follow the regular telemonitoring care pathway, which involves completing the Monitor IBD At Home (MIAH) questionnaire and performing a fecal calprotectin (FCP) home test. The app provides follow-up advice based on the results ofan algorithm. In the on-demand intervention group, patients can use the app at their own discretion when they experience symptoms but are not required to perform standard measurements when they are symptom-free. This allows them to have control over their monitoring activities.

Study population: Adult (>18 years) patients with an established diagnosis of Crohn's disease or ulcerative colitis according to international guidelines, on maintenance therapy with no medication changes in the last three months and in stable remission. Remission will be defined as faecal calprotectin (FCP) < 100 µg/g and Harvey Bradshaw Index (HBI) < 5 for CD and as faecal calprotectin (FCP) < 250 µg/g and Simple Clinical Colitis Activity Index scores (SCCAI) < 3 for UC.

Study parameters/endpoints: Disease activity, defined as the number persistent flares, is the primary outcome measure. The secondary outcome measures include: clinical disease activity (number of flares), patient-reported disease activity (IBD-Control-8), quality of life (EQ-5D-5L, WIX, and SIBDQ), self-efficacy (IBD-SES), patient activation (PAM-13), total number of contacts with a healthcare provider, safety, and costs (healthcare costs, productivity costs, and patient costs). Baseline characteristics include patient, disease, and socio-demographic factors.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years.
* Confirmed IBD diagnosis according to current standards (37).
* Provided informed consent.
* Maintenance therapy with no medication changes in the last 3 months.
* Remission (17, 38)
* Crohn's disease: Faecal calprotectin (FCP) < 100 µg/g and Harvey Bradshaw Index (HBI) < 5 or MIAH-CD < 0.3623618
* Ulcerative Colitis: Faecal calprotectin (FCP) < 250 µg/g and Simple Clinical Colitis Activity Index scores (SCCAI) < 3 or MIAH-CU < 0.354215

Exclusion Criteria:

* Presence of a stoma.
* Presence of an ileo-anal pouch or ileorectal anastomosis.
* Participating in another prospective clinical trial that interferes with this trial.
* Have insufficient knowledge of the Dutch language to use the application.
* Do not have a smartphone or tablet with an internet connection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Persistent Flares | 12 months
  The primary study parameter is the cumulative incidence of persistent flares, defined as a flare for a consecutive period of ≥ 12 weeks during the study period.
  A flare is defined as:
  * The presence of faecal calprotectin more than 250 μg/g on two consecutive FCP-measurements collected at 12 weeks apart and;
  * MIAH score above 0.354215 (ulcerative colitis) or 0.3623618 (Crohn's disease) and least once during the period of 12 weeks.

SECONDARY OUTCOMES:
Number of contacts with healthcare provider | 12 months
  All contacts
Disease activity from patient perspective | 12 months
  Measured with IBD-control 8
Disease activity from clinical perspective as number of flares | 12 months
  Measured with FCP and MIAH
Generic quality of life | 12 months
  Measured with WiX
Generic quality of life and costs | 12 months
  Measured with EQ-5D-5L
Disease specific quality of life | 12 months
  Measured with SIBDQ
Self-efficacy | 12 months
  Measured with IBD-SES
Patient Activation | 12 months
  Measured with PAM-13
Patient safety measured with variables retrieved from the hospital information system | 12 months
  Following variables retrieved from the hospital information system:
  * Number and cumulative length of hospital admissions
  * Number of emergency department visits
  * Number of IBD-related surgeries, distinguish between fistula and non-fistula surgery
  * Cumulative length of corticosteroid usage
  * Mortality
Healthcare costs | 12 months
  Measured with iMCQ
Productivity costs | 12 months
  Measured with iPCQ

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, North Brabant
  - Franciscus, Rotterdam, South Holland

IPD SHARING:
Plan to Share IPD: No